CLINICAL TRIAL: NCT06213753
Title: Complications of Non-Surgical Treatment in Acute Cholecystitis, the Unkonwn Pathway
Brief Title: Complications of Non-Surgical Treatment in Acute Cholecystitis
Status: Completed | Type: Observational
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Ana María González Castillo, Doctor, Hospital del Mar
Other Study IDs: Complications of NST in ACC
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Acute Cholecystitis
Keywords: Acute Cholecystitis; Cholecystectomy; Tokyo Guidelines; Non-Surgical Treatment; Mortality; High-risk patient
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute cholecystitis (AC) is the second most frequent pathology in Surgical Emergencies; laparoscopic cholecystectomy (LC) is the gold standard treatment, but not all patients are fit for surgery. Percutaneous Cholecystostomy (PC) is an alternative to LC but has high comorbidity. There is no protocol in our institution for Non-Surgical Treatment (NST). This study aims to analyse the complications of non-surgical treatment and a new local management algorithm

DETAILED DESCRIPTION:
It's a single-centre retrospective study of 1652 adults with AC from 2011 to 2022, including baseline demographic characteristics, comorbidity severity defined as the Charlson Comorbidity Index (CCI), ASA Score, and Tokyo Guidelines' severity classification. The primary outcome is to study the complications of NST.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of an Acute Cholecystitis.
* Older than 18 years old.

Exclusion Criteria:

* Younger than 18 years old.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients admited with the diagnostic of Acute Cholecystitis
Sampling Method: Non-Probability Sample
Enrollment: 1652 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Complications | 2011-2022
  The main outcome measure was the total of complications in patients with an Acute Calculous Cholecystitis assessed by the Clavien-Dindo Classification.

IPD SHARING:
Plan to Share IPD: No